CLINICAL TRIAL: NCT00500032
Title: Blood Collection for Use in Serological Assay Development From Healthy Adult Volunteers Who Completed Study 6108A1-500
Brief Title: Blood Collection for Use in Serological Assay Development From Healthy Adult Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 6108A1-1000
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Adult
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Active Comparator for all subjects enrolled in 6108A1-500
  Interventions: Procedure: blood draw

INTERVENTIONS:
Procedure: blood draw — Blood draw from subjects previously vaccinated in 6108A1-500 trial

SUMMARY:
Subjects who have completed study 6108A1-500, in which our experimental meningoccal B vaccine or placebo was administered, will be approached for inclusion into this study which is purely for blood draw. The sera will be used for assay development.

DETAILED DESCRIPTION:
The purpose of this protocol is to analyze the collection of blood volumes (approximately 200 to 470 mL per bleed) from volunteer donors who previously completed study 6108A1-500. As such, the inclusion and exclusion criteria are consistent with the Australian Red Cross guidelines for blood donation.

The 6108A1-500 study is an ongoing, double-blind, ascending-dose, randomized, placebo-controlled trial to assess the safety and tolerability of ascending doses of rLP2086 with aluminum phosphate (AlPO4) adjuvant, in healthy adults aged 18 to 25 years. Upon completion of participation in the 6108A1-500 study, subjects will be approached to participate in this blood sampling study. The sites participating in this blood sampling study are the same sites participating in the 6108A1-500 study.

ELIGIBILITY:
Main Inclusion Criteria:

1. Completed study 6108A1-500.
2. Hemoglobin level ≥12.0 and ≤16.5 g/dL for female subjects and ≥13.0 and ≤18.5 g/dL for male subjects.
3. Body weight ≥45 and ≤120 kg.
4. Systolic blood pressure >90 and <180 mm Hg.
5. Diastolic blood pressure >60 and <100 mm Hg.
6. Able to be contacted by telephone.
7. For all female subjects: have a negative urine pregnancy test unless the subject is surgically sterile.

Main Exclusion Criteria:

1. Bleeding diathesis or condition associated with prolonged bleeding time.
2. Prior antibiotic use (within 14 days).
3. Any clinically significant chronic disease that, in the investigator's judgment may be worsened by blood draw.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Primary objective is to obtain blood volumes (approximately 200 to 470 mL per bleed) from volunteer donors who previously completed study 6108A1-500, for use in serological assay development. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Australia: medinfo@wyeth.com
Locations (3):
- Australia (3):
  - Herson, Queensland
  - North Adealaide, South Australia
  - Perth, Western Australia